CLINICAL TRIAL: NCT01108406
Title: Long Term Safety of the Sonitus SoundBite System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonitus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN005.00
Record Dates: First submitted 2010-04-15; First posted 2010-04-22 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Hearing Loss; Unilateral Hearing Loss; Total Unilateral Deafness
Keywords: Hearing Loss; Unilateral Hearing Loss; Single Sided Deafness
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SoundBite Hearing System (Experimental): The objective of this study was to assess the long-term safety and quality of life impact of the SoundBite™ Hearing System.
  Safety was measured in terms of dental, audiological and medical adverse events related to device or procedure.
  Quality of Life was measured in terms of changes in Abbreviated Profile of Hearing Aid Benefit (APHAB) and as reported in a quality of life survey (SSD Questionnaire).
  The duration of the study was 6 months with measures taken at Day 1, 3 months and 6 months.
  Interventions: Device: Sonitus SoundBite System; Device: SoundBite Hearing System

INTERVENTIONS:
Device: Sonitus SoundBite System — Non Surgical Bone Conduction Device
  Other Names: Sonitus Bone Conduction Device
Device: SoundBite Hearing System

SUMMARY:
The objective of this study is to assess the long-term safety and quality of life improvement of the Sonitus SoundBite Hearing System.

DETAILED DESCRIPTION:
The Sonitus Bone Conduction Device (BCD) is a bone conduction device for single-sided deafness (SSD). The Sonitus BCD consists of an Oral Appliance (OA), an external microphone component, worn behind the ear (BTE), a calibration interface cable and a PC-controlled calibration software for subject calibration. The Sonitus BCD picks up sounds from a microphone located within the ear canal of the deaf ear, capitalizing on the acoustics of the natural pinna and ear canal. The signal picked up by the microphone is then transmitted wirelessly to a removeable bone conduction oral appliance located on the upper molars. The oral appliance receives the acoustic signal from the BTE and applies an equivalent vibratory signal to the teeth that reaches the skull via bone conduction and routed transcranially to the contralateral cochlea.

ELIGIBILITY:
Inclusion Criteria:

* Must be >18, <80 years old
* Must be fluent in English, as determined by the PI
* Must not be a member of a vulnerable group (IRB defined)
* Must remain in geographic area during duration of the study
* Diagnosis of acquired SSD (Section 3.1), time since onset (≥3 mos)
* Must have a minimum of 6 posterior teeth remaining in the upper arch (3 teeth per side),third molars are acceptable if healthy, fully erupted and substituting for second molars

Exclusion Criteria:

* Must not be current users of devices such as Baha, CROS or TransEar
* Must not have known active medical causes of SSD

  * Active middle ear pathology
  * Conductive HL (Otosclerosis, otitis media, otitis externa and others)
  * Sudden hearing loss that is not stable
* Must not have known medical problems that might be life-threatening or is a contraindication for elective dental or medical procedures
* Must not have a history of seizures
* Must not have known problems that may interfere with the impression procedure, such as inability to breath through nose (e.g. severe flu, allergies or cold)
* Must not have allergies to polymers
* Must not have known dental abnormalities

  * Temporary crowns or undergoing dental treatment
  * Poor oral hygiene and/or rampant decay
  * Current orthodontics
  * Active caries in one or more of the possible abutment teeth for the device
  * Active moderate to severe periodontal disease around abutment teeth for the device
  * Suspicious oral/facial lesions or swelling of any type
  * Severe pain on palpation on any area of mouth, face or neck
  * Moderate to severe heat sensitivity on any of the upper teeth
  * Subject currently being treated for temporomandibular joint disorder (TMJ), pain, full mouth reconstruction or posterior dental implants
* Must not have known Audiological conditions

  * Conductive hearing loss (air-bone gap >10dB HL at more than 3 frequencies)
  * Word recognition scores inconsistent with pure tone averages
  * Fluctuating hearing loss
* Must not have known psychological factors that interfere with their ability to comply, comprehend, consent and cooperate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Murray, MD, Principal Investigator — Camino ENT
Locations (1):
- Camino Ear Nose and Throat, San Jose, California, United States

REFERENCES:
- [Background] Ozer E, Adelman C, Freeman S, Sohmer H. Bone conduction hearing on the teeth of the lower jaw. J Basic Clin Physiol Pharmacol. 2002;13(2):89-96. doi: 10.1515/jbcpp.2002.13.2.89. PMID 16411423
- [Background] Dahlin GC, Allen FG, Collard EW. Bone-conduction thresholds of human teeth. J Acoust Soc Am. 1973 May;53(5):1434-7. doi: 10.1121/1.1913490. No abstract available. PMID 4712563
- [Background] Wazen JJ, Spitzer J, Ghossaini SN, Kacker A, Zschommler A. Results of the bone-anchored hearing aid in unilateral hearing loss. Laryngoscope. 2001 Jun;111(6):955-8. doi: 10.1097/00005537-200106000-00005. PMID 11404603
- [Background] Wazen JJ, Spitzer JB, Ghossaini SN, Fayad JN, Niparko JK, Cox K, Brackmann DE, Soli SD. Transcranial contralateral cochlear stimulation in unilateral deafness. Otolaryngol Head Neck Surg. 2003 Sep;129(3):248-54. doi: 10.1016/S0194-5998(03)00527-8. PMID 12958575
- [Background] Stenfelt SP, Hakansson BE. Sensitivity to bone-conducted sound: excitation of the mastoid vs the teeth. Scand Audiol. 1999;28(3):190-8. doi: 10.1080/010503999424761. PMID 10489868
- [Background] Moore BC, Popelka GR. Preliminary comparison of bone-anchored hearing instruments and a dental device as treatments for unilateral hearing loss. Int J Audiol. 2013 Oct;52(10):678-86. doi: 10.3109/14992027.2013.809483. Epub 2013 Jul 17. PMID 23859058
- [Background] Murray M, Popelka GR, Miller R. Efficacy and safety of an in-the-mouth bone conduction device for single-sided deafness. Otol Neurotol. 2011 Apr;32(3):437-43. doi: 10.1097/MAO.0b013e3182096b1d. PMID 21221045
- [Background] Miller R, Hujoel P, Murray M, Popelka GR. Safety of an intra-oral hearing device utilizing a split-mouth research design. J Clin Dent. 2011;22(5):159-62. PMID 22403981
- [Background] Popelka GR, Derebery J, Blevins NH, Murray M, Moore BC, Sweetow RW, Wu B, Katsis M. Preliminary evaluation of a novel bone-conduction device for single-sided deafness. Otol Neurotol. 2010 Apr;31(3):492-7. doi: 10.1097/MAO.0b013e3181be6741. PMID 19816229
- [Result] Murray M, Miller R, Hujoel P, Popelka GR. Long-term safety and benefit of a new intraoral device for single-sided deafness. Otol Neurotol. 2011 Oct;32(8):1262-9. doi: 10.1097/MAO.0b013e31822a1cac. PMID 21799455
- See also: product website — http://www.soundbitehearing.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in April 2010. Subjects were informed about the potential for participation via IRB approved flyers or by indicating interest on consent forms from other studies.
Groups:
- Sonitus SoundBite System: Long Term Safety was measured in terms of dental, audiological and medical adverse events related to device or procedure.
Period: Overall Study
Arm/Group | Sonitus SoundBite System
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Long Term Safety: Safety was measured in terms of dental, audiological and medical adverse events related to device or procedure.
Arm/Group | Long Term Safety
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.41 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Long Term Safety
Description: The safety outcomes were defined as no changes in medical, auditory, or dental status and no device or procedure related adverse events during the study period. Safety was evaluated by conducting a Comprehensive Medical evaluation at Enrollment and at study termination; Comprehensive Dental evaluation at Enrollment and at 3 and 6 months, with interim dental checks in between if necessary and Comprehensive Audiological evaluation at Enrollment and at 6 months.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Number of Participants Experiencing no Adverse Events: Safety was measured in terms of dental, audiological and medical adverse events related to device or procedure. Dental measurements included periodontal measurements (bone loss, oral health, bleeding index, calculus, peridontal probing) at baseline compared to 6 months. Audiological included hearing evaluation and aided thresholds baseline compared to 6 months and medical compared medical and ear health baseline compared to 6 months.
Arm/Group | Number of Participants Experiencing no Adverse Events
Number analyzed (Participants) | 22
participants | 22

2. Secondary Outcome: Measurement of Device Benefit With the Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: The measure of the benefit of the device was assessed using the Abbreviated Profile of Hearing Aid Benefit (APHAB) , a 24-item self-assessment inventory in which the amount of difficulty in everyday situations is reported with larger numbers indicating more difficulty. Device benefit is calculated by subtracting the score obtained after using a device from the score obtained before using the device. Software is used to score the APHAB and results are compared from the different timepoints. The APHAB is well characterized and broadly used as a quantifiable measurement. The APHAB benefit scores can range from -99 (treatment worse than no treatment) to +99 (treatment better than no treatment).
Time Frame: 3 months and 6 months
Measure: Mean (Standard Deviation); unit: Global Benefit Score
Groups:
- Global Benefit APHAB Score Aided 3 Months: The Global Benefit APHAB at 3 months endpoint is the change in APHAB scores between the unaided score at the start of the study and the APHAB score after 3 months of therapy.The APHAB Questionnaire produces an overall Global score (GBL). The larger the APHAB benefit score the greater the benefit. A negative APHAB benefit score represents therapy resulting in a worse outcome than no therapy.
- Global Benefit APHAB Score Aided 6 Months: The Global Benefit APHAB at 6 months endpoint is the change in APHAB scores between the unaided score at the start of the study and the APHAB score after 6 months of therapy.The APHAB Questionnaire produces an overall Global score (GBL). The larger the APHAB benefit score the greater the benefit. A negative APHAB benefit score represents therapy resulting in a worse outcome than no therapy.
Arm/Group | Global Benefit APHAB Score Aided 3 Months | Global Benefit APHAB Score Aided 6 Months
Number analyzed (Participants) | 22 | 22
Global Benefit Score | 21.3 (16.9) | 23.1 (16.0)

ADVERSE EVENTS:
Arm/Group | Long Term Safety
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days